CLINICAL TRIAL: NCT00524693
Title: A Double-Blind Placebo Controlled Randomized Trial of Montelukast in Acute Respiratory Syncytial Virus Bronchiolitis
Brief Title: Montelukast in Acute RSV Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Collaborators: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-146-R
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; controlled clinical trial; pediatrics; Infants; montelukast; Respiratory syncytial virus
MeSH Terms: conditions — Bronchiolitis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 4mg Singulair© sachets
  Interventions: Drug: Montelukast
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo granules

INTERVENTIONS:
Drug: Montelukast — 4mg sachets
  Other Names: Singulair©
  Arms: 1
Drug: Placebo granules
  Arms: 2

SUMMARY:
There is evidence of inflammatory mechanisms in RSV bronchiolitis with increased cysteinyl-leukotrienes (cys-LT). Recently, specific cys-LT receptor antagonists - montelukast (Singulair©) approved for use in infants as granule sachets, have become available. We evaluated the effect of Singulair© on clinical progress and on cytokine profiles in the acute phase of RSV bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 4 weeks < 2 years
* Duration of respiratory symptoms < 4 days
* Signs of bronchiolitis: prodromal rhinorrhea and cough, followed by at least two of the following signs: chest retractions, tachypnea, wheezing, or rales
* First episode of wheezing or shortness of breath
* Randomization within 12 hours of admission
* No need for steroid treatment in the ward
* Informed consent

Exclusion Criteria:

* A history of asthma symptoms or any previous hospital admissions with respiratory tract illnesses and if they had ever been treated with anti-asthma medications (prior to the current illness).
* Underlying cardiopulmonary disease such as bronchopulmonary dysplasia, congenital heart disease, immunodeficiency, or cystic fibrosis.

Ages: 4 Weeks to 2 Years | Sex: All
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Length of stay | hours

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, MD, Principal Investigator — Ziv Medical Center

REFERENCES:
- [Derived] Amirav I, Luder AS, Kruger N, Borovitch Y, Babai I, Miron D, Zuker M, Tal G, Mandelberg A. A double-blind, placebo-controlled, randomized trial of montelukast for acute bronchiolitis. Pediatrics. 2008 Dec;122(6):e1249-55. doi: 10.1542/peds.2008-1744. Epub 2008 Nov 4. PMID 18984650